CLINICAL TRIAL: NCT04496453
Title: Development and Testing of ADEPT: A Parent Decision Support for Childhood Vaccinations
Acronym: ADEPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00101904; 1KL2TR002554 (NIH)
Record Dates: First submitted 2020-07-24; First posted 2020-08-03 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Vaccine Refusal
Keywords: childhood vaccines; vaccine hesitancy; vaccination
MeSH Terms: conditions — Vaccination Refusal; Vaccination Hesitancy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Childhood vaccination decision support tool (Experimental): Participants receive childhood vaccination decision support tool
  Interventions: Other: Childhood vaccination decision support tool

INTERVENTIONS:
Other: Childhood vaccination decision support tool — Participants receive childhood vaccination decision support tool

SUMMARY:
The purpose of this study is to develop and evaluate a tool designed to help parents make decisions about childhood vaccines.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Parent or primary caregiver of a child between the ages of 3-6 years who is receiving primary care at Duke.
* Fluent in English

Exclusion Criteria:

* Unable to understand the study objectives, procedures, risks, and benefits
* Unable to consent for themselves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lavanya Vasudevan, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Childhood Vaccination Decision Support Tool
Started | 17
Completed | 11
Not Completed | 6
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | Childhood Vaccination Decision Support Tool
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.06 (7.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Knowledge Related to Childhood Vaccinations as Measured by Study Specific Questionnaire
Description: Study specific questionnaire comprised of 10 True or False questions. Knowledge was measured on a score of 0-10, where a higher score indicates a greater level of knowledge. Outcome reports on the difference in the knowledge score measure pre- and post- exposure to intervention.
Time Frame: pre-survey (baseline) and post-survey (at completion of intervention, approximately 4-6 weeks after baseline)
Population: Participants who completed both questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Childhood Vaccination Decision Support Tool
Number analyzed (Participants) | 11
score on a scale | 1.27 (1.68)

2. Primary Outcome: Change in Acceptability of Childhood Vaccinations
Time Frame: pre-survey (baseline) and post-survey (at completion of intervention, approximately 4-6 weeks after baseline)
Population: Data not collected.
Arm/Group | Childhood Vaccination Decision Support Tool
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Approximately 4-6 weeks
Arm/Group | Childhood Vaccination Decision Support Tool
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT04496453/Prot_SAP_001.pdf
  • Informed Consent Form (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT04496453/ICF_000.pdf